CLINICAL TRIAL: NCT03399760
Title: Evaluation the Dento-alveolar Changes After Platelet Rich Fibrin (i-PRF) Injection During Upper Canine Retraction Using Cone-beam Computed Tomography (CBCT)
Brief Title: Efficacy of Injectable Platelet Rich Fibrin (i-PRF) in Enhancing Bone Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Ortho-01-2018
Record Dates: First submitted 2018-01-08; First posted 2018-01-16 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Malocclusion, Angle Class II, Division 1
Keywords: i-PRF (injectable platelet rich fibrin); alveolar bone height; canine root resorption; bone density; cone-beam computed tomography
MeSH Terms: conditions — Malocclusion, Angle Class II

STUDY DESIGN:
Intervention Model Description: Two Arms injectable platelet rich fibrin group: consisted of two subgroups
  * Experimental group : injectable platelet rich fibrin assisted upper canine retraction
  * Control group: conventional upper canine retraction
Who Masked: Outcomes Assessor
Masking Description: One blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- i-PRF assisted upper canine retraction (Experimental): I-PRF assisted upper canine retraction will be performed in one side of patients with Class II Division 1 malocclusion patients requiring therapeutic extraction of the maxillary first premolars
  Interventions: Biological: i-PRF; Procedure: canine retraction
- conventional upper canine retraction (Experimental): Conventional upper canine retraction will be performed in the other side of patients with Class II Division 1 malocclusion patients requiring therapeutic extraction of the maxillary first premolars
  Interventions: Procedure: canine retraction

INTERVENTIONS:
Biological: i-PRF — i-PRF (injectable platelet rich fibrin) assisted upper canine retraction
  Arms: i-PRF assisted upper canine retraction
Procedure: canine retraction — upper canine retraction will be performed in one side of patients with Class II Division 1 malocclusion patients requiring therapeutic extraction of the maxillary first premolars

SUMMARY:
Twenty patients need therapeutic extraction of the maxillary first premolars with subsequent retraction of the maxillary canines, will be divided randomly into two groups, and will randomly assigned to one side of the maxillary arch at the first premolar region, and the other side served as the control. Canine retraction will be initiated after completion of the leveling and alignment phase via closed nickel-titanium coil springs applying 150 g of force per side. Soldered transpalatal arch will be used as an anchor unit. The dento-alveolar changes will be assessed immediately before retraction and after 6 months using CBCT.

DETAILED DESCRIPTION:
Extraction is a procedure that is currently performed in orthodontics, either in the context of early treatment or for adolescents with severe crowding or protrusion/overjet. The consequences of this ''simple'' procedure may show up many mucosal and osseous complications such as: bone resorption with collapse of the alveolar process, a gingival cleft or gingival recession in the area surrounding the extraction site. Besides the potential esthetic repercussions, these periodontal defects also give rise to a clinical problem with achieving some orthodontic movements, such as complete closure of the space or uprighting a root.

A systematic review evaluating alveolar bone dimension changes of extraction sockets showed a range of width reduction of 2.6-4.6mm, Two-thirds of the loss occurred in the first 3 months, the remodeling of alveolar bone in the extraction site always decreases ridge volume and deforms the ridge configuration which impairs orthodontic movement of the tooth posteriorly.

Endogenously produced biologicals have been tested based on their roles in the turnover of alveolar bone in response to orthodontic tooth movement as well as during wound healing.

From here it has been thought about using a method to enhance bone quality after extraction. The platelet rich fibrin (PRF) has the ability to enhance tissue regeneration, accelerate wound healing and inducing stem cells differentiation through its growth factors (GFs).

PRF characteristics in comparison to platelet rich plasma PRP are:

1. its preparation is completely natural and there is no need for thrombin addition so there isn't immune reaction
2. it contains stem cells
3. it requires one stage centrifugation
4. PRF has been reported to gradually release autologous growth factors and expressed stronger and more durable effect on the cellular proliferation and differentiation than PRP in vitro This is the first study in the world that will use i-PRF with Orthodontic treatment, because of its benefits and easiness of using in dental clinic Study sample that consists of 20 patients, Allocation of the sides of intervention (PRF injection) and control sides is made by computer program (Excel).

After ensuring of the patients compliance with the terms and conditions of this study, the purpose and methods of the study will be explained to the patients using Information Sheet. In case of approval to participate, the patients asked to sign the Informed Consent.

Extra & Intra-oral photographs, impressions and clinical examination will be made.

Canine retraction will be initiated after completion of the leveling and alignment phase via closed nickel-titanium coil springs applying 150 g of force per side at the same time 20ml of patients' blood will be withdrawn and centrifuged (700 rpm within 3 minutes) to get 4ml i-PRF. PRF will be injected at the area of the extracted first premolar, The first point place is in the buccal interventional side (supra periosteal injection) and the second point place is in the palatal interventional side(sub periosteal injection). PRF will be injected twice at the beginning and at the middle of the canine retraction.

High resolution CBCT will be taken before the beginning of canine retraction (T0) and after 6 months (T1).

ELIGIBILITY:
Inclusion Criteria:

1. Adult healthy patients, Male and female, Age range: 15-27 years.
2. Class II Division 1 malocclusion:

   * Mild / moderate skeletal Class II (ANB ≤7)
   * Overjet ≤10
   * Normal or excessive facial height (Clinically and then cephalometry assessed using these angles : SN-MP , MM , Y axis)
   * Mild to moderate crowding ≤ 4
3. permanent occlusion.
4. Exist all the upper teeth (except third molars).
5. Good oral and periodontal health:

   * Probing depth < 4 mm
   * No radiographic evidence of bone loss.
   * Gingival index ≤ 1
   * Plaque index ≤ 1

Exclusion Criteria:

1. Medical problems that affect tooth movement (corticosteroid, NSAIDs, …)
2. patients have anti indication for oral surgery ( medical - social - psycho)
3. Presence of primary teeth in the maxillary arch
4. Missing permanent maxillary teeth (except third molars).
5. Poor oral hygiene or Current periodontal disease:

   * Probing depth ≥ 4 mm
   * radiographic evidence of bone loss
   * Gingival index > 1
   * Plaque index > 1
6. Patient had previous orthodontic treatment
7. Craniofacial anomalies (cleft lip and palate patients)
8. Smokers
9. coagulation disorders and patients treated with anticoagulants.
10. patients with immunodeficiency disorders

Ages: 15 Years to 27 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2017-08-20 (Actual); Primary Completion 2019-01-20 (Actual); Study Completion 2019-07-10 (Actual)

PRIMARY OUTCOMES:
Canine root resorption | After 6 months from the beginning of canine retraction
  Root length measurement from a reference line between buccal and palatal cemento-enamel junction (CEJ) to apex. These lines are perpendicular to the long axis of the canine. The levels of CEJ and root apex were assessed using a combination of axial, sagittal, and coronal images.

SECONDARY OUTCOMES:
Alveolar bone height in the first premolar region | After 6 months from the beginning of canine retraction
  By measuring the distance between two lines:
  The first line: the line passing through the distal and mesial cemento-enamel junction of the canine The second line: the line passing through the crest of the alveolus distal to the canine
Bone density | After 6 months from the beginning of canine retraction
  By using Hounsfield Unites (Gray Values)

CONTACTS AND LOCATIONS:
Overall Officials: Rania Haddad, PhD., Study Director — Department of Orthodontics, Faculty of Dentistry, Damascus University, Damascus, Syria
Locations (1):
- Damascus University, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No
The Individual participant data will be only available for the researchers in the department of Orthodontics, Damascus University

REFERENCES:
- [Background] Malmgren O, Goldson L, Hill C, Orwin A, Petrini L, Lundberg M. Root resorption after orthodontic treatment of traumatized teeth. Am J Orthod. 1982 Dec;82(6):487-91. doi: 10.1016/0002-9416(82)90317-7. PMID 6961819
- [Background] Lund H, Grondahl K, Grondahl HG. Cone beam computed tomography for assessment of root length and marginal bone level during orthodontic treatment. Angle Orthod. 2010 May;80(3):466-73. doi: 10.2319/072909-427.1. PMID 20050738
- [Background] Dohan Ehrenfest DM, de Peppo GM, Doglioli P, Sammartino G. Slow release of growth factors and thrombospondin-1 in Choukroun's platelet-rich fibrin (PRF): a gold standard to achieve for all surgical platelet concentrates technologies. Growth Factors. 2009 Feb;27(1):63-9. doi: 10.1080/08977190802636713. PMID 19089687
- [Background] Naik B, Karunakar P, Jayadev M, Marshal VR. Role of Platelet rich fibrin in wound healing: A critical review. J Conserv Dent. 2013 Jul;16(4):284-93. doi: 10.4103/0972-0707.114344. PMID 23956527
- [Background] Van der Weijden F, Dell'Acqua F, Slot DE. Alveolar bone dimensional changes of post-extraction sockets in humans: a systematic review. J Clin Periodontol. 2009 Dec;36(12):1048-58. doi: 10.1111/j.1600-051X.2009.01482.x. PMID 19929956
- [Derived] Zeitounlouian TS, Zeno KG, Brad BA, Haddad RA. Three-dimensional evaluation of the effects of injectable platelet rich fibrin (i-PRF) on alveolar bone and root length during orthodontic treatment: a randomized split mouth trial. BMC Oral Health. 2021 Mar 2;21(1):92. doi: 10.1186/s12903-021-01456-9. PMID 33653326